CLINICAL TRIAL: NCT02851914
Title: An Open-Label Pilot Study Comparing the Efficacy of Selective Serotonin Re-Uptake Inhibitors (SSRIs) Versus Tricyclic Antidepressants (TCAs) for Treating Depression in Amyotrophic Lateral Sclerosis
Brief Title: SSRIs vs. TCAs for Depression in ALS Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Ghazala Hayat, Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22974
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Depression; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Depression; Amyotrophic Lateral Sclerosis | interventions — Antidepressive Agents, Tricyclic; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - TCA (Active Comparator): The Tricyclic Antidepressant ("TCA") group will receive medication for 12 weeks. Patients will be evaluated every 4 weeks and phone call will be made in between visits to assess the effectiveness and side effects of the medication. Questionnaires will be repeated in the clinic visits and will be used in the data analysis to look for improvements and to compare the two classes of medication in this study.
  Interventions: Drug: Tricyclic Antidepressants ("TCA")
- Arm 2 - SSRI (Active Comparator): The Selective Serotonin Reuptake Inhibitor ("SSRI") group will receive medication for 12 weeks. Patients will be evaluated every 4 weeks and phone call will be made in between visits to assess the effectiveness and side effects of the medication. Questionnaires will be repeated in the clinic visits and will be used in the data analysis to look for improvements and to compare the two classes of medication in this study.
  Interventions: Drug: Selective Serotonin Uptake Inhibitors ("SSRI")

INTERVENTIONS:
Drug: Tricyclic Antidepressants ("TCA") — if patient shows signs of depression they will be placed on one of these medications and seen by a psychiatrist.
  Arms: Arm 1 - TCA
Drug: Selective Serotonin Uptake Inhibitors ("SSRI") — if patient shows signs of depression they will be placed on one of these medications and seen by a psychiatrist.
  Arms: Arm 2 - SSRI

SUMMARY:
Depression is seen in 9-11% of ALS patients and adequate and proper treatment is needed. In this study, ALS patients will be screened for depression using self-reported multiple choice questionnaire. Patients who fulfill the criteria for depression based on this screening tool will be evaluated by psychiatrist before inclusion in the study. The investigators will also measure quality of life and functional status by simple questionnaires. The patients will be allocated into two treatment groups to receive either TCA or SSRI for 12 weeks. Patients will be evaluated every 4 weeks and phone calls will be made in between the visits if needed to assess about efficacy and any side effects. If any patient reports having suicidal thoughts on any of these phone calls or clinic visits, he/she will be immediately sent to the ER for appropriate management. The investigators will repeat the questionnaires in the clinic visits, and use them in the data analysis to look for any improvement and to compare the two medication classes used in this study. This data may be used later on to do larger studies and help to make standard recommendations in treating depression in ALS patients.

DETAILED DESCRIPTION:
This study is a 12-week, open-label, non-randomized, pilot clinical intervention trial. This is investigator initiated study.This trial will be done at St Louis University ALS clinic. ALS patients will be screened for depression using Beck depression inventory (BDI-II) scale. A mental healthcare provider will evaluate the patients scoring 19 or above, before inclusion in the study. Quality of Life (QOL) assessment by questionnaire (McGill) and ALS functional rating scale (ALS-FRS) measurement will be done at the baseline. Then these patients will be allocated into two treatment groups to receive either TCA or SSRI medication for 12 weeks based on the clinical judgment (non-randomized). Patients will require clinical encounters every 4 weeks and telephone encounters in between the visits to assess the effectiveness of medication and tolerability of the side effects if any. If any patient endorses active suicidal ideation on any of these assessments, he/she will be immediately sent to the ER for appropriate management. At 4, 8 and 12-week clinic visits, repeat BDI, QOL and ALS-FRS measurement will be done on each patient from both groups and used in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of definite or probable ALS
* Informed and written consent for enrollment in study
* Gender: both male and female
* Age: 25-80 years
* BDI score 19 or above
* Depression diagnosis by mental health provider

Exclusion Criteria:

* History of psychotic disorder, premorbid bipolar depression
* ALS-FRS score < 26
* Cognitive impairment
* Currently on SSRIs or TCAs. However if for some reason they are off their treatment, then they can be enrolled in the study after a washout period of 30 days.
* Currently on other antidepressants such as monoamine oxidase inhibitors (MAOIs), selective norepinephrine re-uptake inhibitors (SNRIs) etc.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
BDI-II | Baseline to 12 weeks
  Primary outcome parameter will be relative change in BDI-II score from baseline to 12 weeks

SECONDARY OUTCOMES:
ANCOVA | 12 weeks
  Analysis of covariance will be used to evaluate for significant differences in BDI-II mean scores between the two treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Sean E Goretzke, MD, Study Chair — St. Louis University
Locations (1):
- Monteleone Hall, Saint Louis University, 1438 South Grand Blvd., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No